CLINICAL TRIAL: NCT01697839
Title: Correlation Between Serum Vitamin D Levels and the Incidence of Peripheral Neuropathy Among Multiple Myeloma Patients Who Have Previously Received Treatment With Bortezomib or Thalidomide
Brief Title: Serum Vitamin D Levels and Peripheral Neuropathy Among Multiple Myeloma Patients
Status: Completed | Type: Observational
Sponsor: Oncotherapeutics (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: X05392
Record Dates: First submitted 2012-08-24; First posted 2012-10-02 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma; Peripheral Neuropathy
MeSH Terms: conditions — Multiple Myeloma; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, white blood cells, red blood cells
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective study investigating the relationship between vitamin D and peripheral neuropathy (PN) among multiple myeloma (MM) patients treated with either bortezomib or thalidomide. The study consists of a screening period of up to 14 days, followed by a single assessment visit to evaluate vitamin D levels, incidence and severity of PN, neuropathic pain, and markers of depression. Patient charts will also be utilized to assess the frequency of skeletal-related events.

DETAILED DESCRIPTION:
Approximately 10% of myeloma patients present at diagnosis with clinical neuropathy although studies reveal as many as 1/3 may have abnormal electrophysiological examinations. Baseline neuropathic abnormal findings are exacerbated by many myeloma treatments, especially bortezomib, thalidomide, and to a lesser extent lenalidomide. Several studies suggest that vitamin D supplementation may help reduce the symptoms of neuropathy.In this prospective study, we will investigate the relationship between vitamin D and PN among MM patients treated with either bortezomib or thalidomide. The study consists of a screening period of up to 14 days, followed by a single assessment visit to evaluate vitamin D levels, incidence and severity of PN, neuropathic pain, and markers of depression. Patient charts will also be utilized to assess the frequency of skeletal-related events.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Prior diagnosis of multiple myeloma based on standard criteria (Durie 1986)
* Received consecutive, prior treatment for MM with a regimen consisting of at least 16 consecutive weeks of bortezomib or 16 consecutive weeks of thalidomide prior to the Day of Assessment
* The 16 weeks of consecutive treatment must have included at least one of the following doses and schedules:

  * Bortezomib: ≥ 1.0 mg/m² dosed 3 or more times per each 4-week period
  * Thalidomide: ≥ 50 mg/day dosed daily
* The qualifying regimen may include both bortezomib and thalidomide. However, the above inclusion requirements need only be satisfied by either one of the agents.
* Age ≥18 years at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes (POEMS) syndrome (Bardwick 1980)
* Plasma cell leukemia
* Primary amyloidosis
* Vitamin D level assessment occurring within the 12 months preceding the Day of Assessment
* Vitamin D non-dietary oral supplementation > 1200 IU per day for > 30 total days within the 12 month period preceding the Day of Assessment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D levels | Day 1
  Correlation of serum vitamin D levels to the incidence and severity of anti-myeloma treatment-induced PN/ neuropathic pain among MM patients previously exposed to bortezomib and/or thalidomide

SECONDARY OUTCOMES:
Skeletal related event | Day 1
  Correlation between vitamin D levels and skeletal-related events (pathologic fracture, spinal cord compression or collapse, or surgery or radiotherapy to bone) among MM patients

OTHER OUTCOMES:
Markers of depression | Day 1
  Correlation between vitamin D levels and markers of depression for MM patients

CONTACTS AND LOCATIONS:
Overall Officials: James R. Berenson, M.D., Principal Investigator — Oncotherapeutics
Locations (3):
- United States (3):
  - Beaver Medical Group, Highland, California
  - James R. Berenson M.D., Inc., West Hollywood, California
  - Illinois Cancer Specialists, Hinsdale, Illinois